CLINICAL TRIAL: NCT01947842
Title: Effect of a Smartphone Application on Oral Contraceptive Adherence in College Females: a Randomized-controlled Trial.
Brief Title: Effect of a Smartphone Application on Oral Contraceptive Adherence in College Females
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding unavailable.
Sponsor: Belmont University (Other)
Responsible Party: Principal Investigator, Adam Pace, Assistant Professor of Pharmacy Practice, Belmont University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BUCOP-001
Record Dates: First submitted 2013-09-18; First posted 2013-09-23 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Adherence to Oral Contraceptive Therapy
Keywords: Smartphone; adherence; contraceptives; college; females

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smartphone App (Experimental): The pharmacist will download and configure the Dosecast smartphone application to remind the patient to take their medication in addition to pharmacist counseling on the importance of adherence.
  Interventions: Device: Smartphone App Dosecast
- Counseling Alone (No Intervention): This arm will receive only counseling from the pharmacist with no other intervention.

INTERVENTIONS:
Device: Smartphone App Dosecast — The Dosecast app is configured to remind the patient to take their medication.
  Arms: Smartphone App

SUMMARY:
This research study is to see if smartphone applications help college women remember to take birth control better than pharmacist consultation alone. Patients will participate in this study for 6 (six) months. The study will have two groups. Patients will be randomly assigned to one group or the other. The control group will be counseled by the pharmacist on the importance of taking birth control as prescribed. The study group will get the same counseling, but will also be set up to receive reminders to take medication on a smartphone application called Dosecast.

ELIGIBILITY:
Inclusion Criteria:

* female gender
* 18-29 years of age
* current prescription for an OCP
* currently enrolled as a student at the institution associated with the pharmacy
* possession of a compatible smartphone.

Exclusion Criteria:

* Pregnant patients
* Patients who become pregnant during the study will discontinue, but their data up until time of discontinuation will be used
* Patients using other forms of contraception (patch, injection, IUD, intra-vaginal ring, implant).

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Doses Missed | 6 months
  Number of doses of oral contraceptive missed over a six-month period.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Auburn University, Auburn, Alabama
  - University of Mississippi, Oxford, Mississippi
  - Belmont University, Nashville, Tennessee